CLINICAL TRIAL: NCT06067451
Title: Impact of SMART GOAL Setting Protocol on Body Weight and Metabolic Parameters in Children and Adolescents With Prediabetes; a Randomized Clinical Trial.
Brief Title: SMART GOALS for Youth With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-0375
Record Dates: First submitted 2023-09-15; First posted 2023-10-04 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: PreDiabetes; Adolescent Obesity; Behavior, Health; Nutritional and Metabolic Diseases; Diet Habit; Lifestyle Risk Reduction
Keywords: Nutrition
MeSH Terms: conditions — Prediabetic State; Pediatric Obesity; Health Behavior; Nutritional and Metabolic Diseases; Feeding Behavior; Risk Reduction Behavior | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: We'll enroll 60 pediatric subjects diagnosed with prediabetes within three months at the Pediatric Diabetes Clinic. These subjects will be randomly assigned to two arms. All participants will receive standardized medical nutrition therapy protocol and visit frequency from RD. Study group participants will get the SGSP, consisting of the SMART Goal Selection Guide (SGSG) and Weekly Goal Monitoring Tool (WGMT). SGSG will outline three SMART goal domains (exercise, diet, behavior) with a primary goal and example goals. Participants will personalize 2-3 SMART goals, those in standard of care group will just be asked "what changes they plan to make".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART GOAL Arm (Experimental): The participants randomized to the study group will receive the SGSP, consisting of the SMART Goal Selection Guide (SGSG) and Weekly Goal Monitoring Tool (WGMT), which will be used in tandem.
  The study group participants will also be asked to summarize the information discussed during the visit, and then will receive the SMART (Specific, Measurable, Attainable, Realistic, Time sensitive) Goal Setting Protocol (SGSP).
  Interventions: Behavioral: SMART GOALS Setting Tool/ Protocol
- Standard of Care Arm (No Intervention): Participants randomized to this group will receive standard of care.
  At the end of each visit, the participants in the standard of care (SOC) group will be asked to provide a summary of topics discussed and what they plan to improve on from now and their next visit:

INTERVENTIONS:
Behavioral: SMART GOALS Setting Tool/ Protocol — The participants randomized to the study group will receive the SGSP, consisting of the SMART Goal Selection Guide (SGSG) and Weekly Goal Monitoring Tool (WGMT), which will be used in tandem. The participant will first receive the SGSG which will highlight 3 domains of SMART goals (exercise, diet, and behavior). Each domain will have 1 predetermined and unchanging primary goal which will serve as the standard for all participants to strive for.
  Arms: SMART GOAL Arm

SUMMARY:
The goal of this study is to compare the impact of a SMART ((specific, measurable, attainable, realistic, or timely) Goal setting protocol on body weight, metabolic parameters (Hemoglobin A1c, lipids), diet quality and physical activity frequency in obese children with prediabetes in the outpatient setting. The main question is if participants using the SMART Goal Setting Protocol (SGSP) will have a significant reduction. The participants randomized to the study group will receive the SGSP, consisting of the SMART Goal Selection Guide (SGSG) and Weekly Goal Monitoring Tool (WGMT), in BMI Z-score, A1c, and dyslipidemia in 6 months compared to controls.

DETAILED DESCRIPTION:
Implementing a SMART goal-setting protocol for the overweight and obese pediatric population with prediabetes can benefit patients by empowering participants to set their own goals. In addition, utilizing a standardized tool can provide a more focused approach to behavior change between visits and increase a child's sense of self- efficacy and autonomy which may enhance motivation and engagement in the treatment process. This study can add strength to current interventions involving childhood obesity and prediabetes management and may inform the development of a more effective interventions in this population. By providing evidenced-based strategies, this study has the potential to improve the health of children at risk for type 2 diabetes.

The investigators will recruit 60 participants with newly diagnosed prediabetes to the proposed study.

Participants will be recruited from the outpatient clinic of the Children's Diabetes Center at the Cohen Children's Medical Center, Long Island, NY.

Participants will be randomized in a 1:1 ratio to one of the two arms. The participants will be stratified by Tanner stage (II and III vs IV and V) and sex (Male vs Female) before randomization.

The Medical Nutrition therapy (MNT) Protocol and visit frequency will be the same for all of the study participants in both the study and standard of care group in which the Registered Dietician (RD) will reinforce and encourage healthy habits and behaviors In addition successes and barriers to change.

At the end of each visit, the participants in the standard of care (SOC) group will be asked to provide a summary of topics discussed and what the participants plan to improve on from now and their next visit: responses will be documented in the EMR, and participants will schedule a follow-up visit in 1-4 months.

The participant randomized in the study group will first receive the SGSG which will highlight 3 domains of SMART goals (exercise, diet, and behavior). Each domain will have 1 predetermined and unchanging primary goal which will serve as the standard for all participants to strive for based on the latest literature recommendations. In addition, each domain will provide a list of examples of SMART goals for participants to choose from. Participants will be asked to independently select and personalize 2-3 SMART goals from this list.

The Registered Dietitian will identify the patient's perceived challenges in achieving their goal, work collaboratively with the patient to problem-solve and make necessary modifications to the goal to overcome challenges. The provider may suggest scaling back the goal if participant reports that perceived challenges are deemed to be significant or participants may choose to work on new goals or will intensify current goals as necessary at the end of each follow-up. The goal will be recorded in the WGMT for progress evaluation and monitoring. This tool should be returned at follow-up. The WGMT will be documented into the patients' chart and scanned into the Electronic Medical Record (EMR).

The study will evaluate changes in weight throughout the intervention by measuring participants anthropometric parameters, including height, weight, and BMI. These measurements will be taken at baseline, 1-4 months, and 4-7 months using the Touchbase Electronic medical record system, which will calculate BMI based on CDC growth charts adjusted for age and sex based.

To assess changes in metabolic parameters, routine laboratory data will be collected based on the discretion of the attending endocrinologist per the standard of care. This will include Hemoglobin A1c, lipid panel and blood pressure. The data will be used to evaluate changes in metabolic health over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Children between ages 10-18 years at baseline visit
2. Children with BMI for age and sex ≥ 85th percentile at baseline visit
3. Children with hemoglobin A1c 5.7% to 6.4% at baseline visit

Exclusion Criteria:

1. Children who are not able to provide assent to the study
2. Children less than 10 years in age
3. Children that are not interested in weight loss or diet and lifestyle change
4. Children with known diabetes that use medications that alter glucose or lipid metabolism such as (insulin, metformin, Glucagon Like Peptide-1 Receptor Antagonist (GLP-1 RA), Statins, Accutane).
5. Children on medications that can alter body weight (including antidepressants, steroids, stimulants).
6. Children with documented learning and/or intellectual disabilities as identified through the electronic medical record (such as cognitive disability or autism spectrum disorder)
7. Children with known psychiatric disorders disabilities as identified through the electronic medical record (e.g., schizophrenia, depression, bipolar disorder, or psychosis
8. Children that have known medical conditions, including endocrine dysfunction, Cushing's Syndrome, or other systemic illness
9. Children with known or suspected eating disorders as identified through the electronic medical record
10. Children that have known genetic or syndromic obesity
11. Female children who are pregnant

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of SMART Goal setting on BMI z-scores To determine the impact of SMART Goal setting on BMI z-scores | 6 months
  To determine the impact of SMART Goal setting on BMI z-scores, will assess anthropometrics at baseline, month 3 and at final visit (month 6)

SECONDARY OUTCOMES:
Temporal changes in Hemoglobin A1c between the study and control groups | 3 months
  A1c will be drawn every 3 months.
Temporal changes in Lipids | 6 months
  Lipid panel to be drawn at baseline and again at 6 months if show elevation are detected per standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U. Nwosu, MD, Principal Investigator — NORTHWELL HEALTH, INC.
Locations (1):
- Northwell Health, New York, New York, United States

REFERENCES:
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Flechtner-Mors M, Thamm M, Wiegand S, Reinehr T, Schwab KO, Kiess W, Widhalm K, Holl RW; APV initiative and the BMBF Competence Network Obesity. Comorbidities related to BMI category in children and adolescents: German/Austrian/Swiss Obesity Register APV compared to the German KiGGS Study. Horm Res Paediatr. 2012;77(1):19-26. doi: 10.1159/000334147. Epub 2011 Nov 22. PMID 22104037
- [Background] Han JC, Lawlor DA, Kimm SY. Childhood obesity. Lancet. 2010 May 15;375(9727):1737-48. doi: 10.1016/S0140-6736(10)60171-7. Epub 2010 May 5. PMID 20451244
- [Background] Daniels SR. Complications of obesity in children and adolescents. Int J Obes (Lond). 2009 Apr;33 Suppl 1:S60-5. doi: 10.1038/ijo.2009.20. PMID 19363511
- [Background] Wing RR, Lang W, Wadden TA, Safford M, Knowler WC, Bertoni AG, Hill JO, Brancati FL, Peters A, Wagenknecht L; Look AHEAD Research Group. Benefits of modest weight loss in improving cardiovascular risk factors in overweight and obese individuals with type 2 diabetes. Diabetes Care. 2011 Jul;34(7):1481-6. doi: 10.2337/dc10-2415. Epub 2011 May 18. PMID 21593294
- [Background] Weiss R, Taksali SE, Tamborlane WV, Burgert TS, Savoye M, Caprio S. Predictors of changes in glucose tolerance status in obese youth. Diabetes Care. 2005 Apr;28(4):902-9. doi: 10.2337/diacare.28.4.902. PMID 15793193
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Kelley CP, Sbrocco G, Sbrocco T. Behavioral Modification for the Management of Obesity. Prim Care. 2016 Mar;43(1):159-75, x. doi: 10.1016/j.pop.2015.10.004. PMID 26896208
- [Background] International Pediatric Endosurgery Group (IPEG). IPEG guidelines for surgical treatment of extremely obese adolescents. J Laparoendosc Adv Surg Tech A. 2009 Apr;19 Suppl 1:xiv-xvi. doi: 10.1089/lap.2009.9981.supp. No abstract available. PMID 19371154
- [Background] Armstrong SC, Bolling CF, Michalsky MP, Reichard KW; SECTION ON OBESITY, SECTION ON SURGERY. Pediatric Metabolic and Bariatric Surgery: Evidence, Barriers, and Best Practices. Pediatrics. 2019 Dec;144(6):e20193223. doi: 10.1542/peds.2019-3223. Epub 2019 Oct 27. PMID 31656225
- [Background] Ameer B, Weintraub MA. Pediatric Obesity: Influence on Drug Dosing and Therapeutics. J Clin Pharmacol. 2018 Oct;58 Suppl 10:S94-S107. doi: 10.1002/jcph.1092. PMID 30248198
- [Background] Williams CF, Bustamante EE, Waller JL, Davis CL. Exercise effects on quality of life, mood, and self-worth in overweight children: the SMART randomized controlled trial. Transl Behav Med. 2019 May 16;9(3):451-459. doi: 10.1093/tbm/ibz015. PMID 31094443
- [Background] Styne DM, Arslanian SA, Connor EL, Farooqi IS, Murad MH, Silverstein JH, Yanovski JA. Pediatric Obesity-Assessment, Treatment, and Prevention: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2017 Mar 1;102(3):709-757. doi: 10.1210/jc.2016-2573. PMID 28359099
- [Background] Al-Khudairy L, Loveman E, Colquitt JL, Mead E, Johnson RE, Fraser H, Olajide J, Murphy M, Velho RM, O'Malley C, Azevedo LB, Ells LJ, Metzendorf MI, Rees K. Diet, physical activity and behavioural interventions for the treatment of overweight or obese adolescents aged 12 to 17 years. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD012691. doi: 10.1002/14651858.CD012691. PMID 28639320
- [Background] Gallo S, Cheskin LJ. Treatment of Obesity: Beyond the Diet. Gastroenterol Clin North Am. 2021 Mar;50(1):113-125. doi: 10.1016/j.gtc.2020.10.003. Epub 2021 Jan 5. PMID 33518158
- [Background] Whitehead L, Glass CC, Abel SL, Sharp K, Coppell KJ. Exploring the role of goal setting in weight loss for adults recently diagnosed with pre-diabetes. BMC Nurs. 2020 Jul 15;19:67. doi: 10.1186/s12912-020-00462-6. eCollection 2020. PMID 32684841
- [Background] Saelens BE, Sallis JF, Wilfley DE, Patrick K, Cella JA, Buchta R. Behavioral weight control for overweight adolescents initiated in primary care. Obes Res. 2002 Jan;10(1):22-32. doi: 10.1038/oby.2002.4. PMID 11786598
- [Background] Liu X, Hanseman DJ, Champagne CM, Bray GA, Qi L, Williamson DA, Anton SD, Sacks FM, Tong J. Predicting Weight Loss Using Psychological and Behavioral Factors: The POUNDS LOST Trial. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1274-83. doi: 10.1210/clinem/dgz236. PMID 31802116
- [Background] Lawrence JM, Divers J, Isom S, Saydah S, Imperatore G, Pihoker C, Marcovina SM, Mayer-Davis EJ, Hamman RF, Dolan L, Dabelea D, Pettitt DJ, Liese AD; SEARCH for Diabetes in Youth Study Group. Trends in Prevalence of Type 1 and Type 2 Diabetes in Children and Adolescents in the US, 2001-2017. JAMA. 2021 Aug 24;326(8):717-727. doi: 10.1001/jama.2021.11165. PMID 34427600
- [Background] Magge SN, Silverstein J, Elder D, Nadeau K, Hannon TS. Evaluation and Treatment of Prediabetes in Youth. J Pediatr. 2020 Apr;219:11-22. doi: 10.1016/j.jpeds.2019.12.061. Epub 2020 Mar 3. No abstract available. PMID 32143933
- [Background] Wallace AS, Wang D, Shin JI, Selvin E. Screening and Diagnosis of Prediabetes and Diabetes in US Children and Adolescents. Pediatrics. 2020 Sep;146(3):e20200265. doi: 10.1542/peds.2020-0265. Epub 2020 Aug 10. PMID 32778539
- [Background] Smith JD, Fu E, Kobayashi MA. Prevention and Management of Childhood Obesity and Its Psychological and Health Comorbidities. Annu Rev Clin Psychol. 2020 May 7;16:351-378. doi: 10.1146/annurev-clinpsy-100219-060201. Epub 2020 Feb 25. PMID 32097572
- [Background] Bendor CD, Bardugo A, Pinhas-Hamiel O, Afek A, Twig G. Cardiovascular morbidity, diabetes and cancer risk among children and adolescents with severe obesity. Cardiovasc Diabetol. 2020 Jun 13;19(1):79. doi: 10.1186/s12933-020-01052-1. PMID 32534575
- [Background] Rupp K, McCoy SM. Bullying Perpetration and Victimization among Adolescents with Overweight and Obesity in a Nationally Representative Sample. Child Obes. 2019 Jul;15(5):323-330. doi: 10.1089/chi.2018.0233. Epub 2019 May 7. PMID 31062988
- [Background] Fryar CD, Kruszon-Moran D, Gu Q, Ogden CL. Mean Body Weight, Height, Waist Circumference, and Body Mass Index Among Adults: United States, 1999-2000 Through 2015-2016. Natl Health Stat Report. 2018 Dec;(122):1-16. PMID 30707668
- [Background] Khera AV, Chaffin M, Wade KH, Zahid S, Brancale J, Xia R, Distefano M, Senol-Cosar O, Haas ME, Bick A, Aragam KG, Lander ES, Smith GD, Mason-Suares H, Fornage M, Lebo M, Timpson NJ, Kaplan LM, Kathiresan S. Polygenic Prediction of Weight and Obesity Trajectories from Birth to Adulthood. Cell. 2019 Apr 18;177(3):587-596.e9. doi: 10.1016/j.cell.2019.03.028. PMID 31002795
- [Background] Hoyt LT, Kushi LH, Leung CW, Nickleach DC, Adler N, Laraia BA, Hiatt RA, Yen IH. Neighborhood influences on girls' obesity risk across the transition to adolescence. Pediatrics. 2014 Nov;134(5):942-9. doi: 10.1542/peds.2014-1286. Epub 2014 Oct 13. PMID 25311606
- [Background] Hu EY, Ramachandran S, Bhattacharya K, Nunna S. Obesity Among High School Students in the United States: Risk Factors and Their Population Attributable Fraction. Prev Chronic Dis. 2018 Nov 8;15:E137. doi: 10.5888/pcd15.180122. PMID 30412690
- [Background] Akinbami LJ, Chen TC, Davy O, Ogden CL, Fink S, Clark J, Riddles MK, Mohadjer LK. National Health and Nutrition Examination Survey, 2017-March 2020 Prepandemic File: Sample Design, Estimation, and Analytic Guidelines. Vital Health Stat 1. 2022 May;(190):1-36. PMID 35593699
- [Background] Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of Obesity and Severe Obesity in US Children, 1999-2016. Pediatrics. 2018 Mar;141(3):e20173459. doi: 10.1542/peds.2017-3459. PMID 29483202
- [Background] The NS, Suchindran C, North KE, Popkin BM, Gordon-Larsen P. Association of adolescent obesity with risk of severe obesity in adulthood. JAMA. 2010 Nov 10;304(18):2042-7. doi: 10.1001/jama.2010.1635. PMID 21063014
- [Background] Wang Y, Beydoun MA, Min J, Xue H, Kaminsky LA, Cheskin LJ. Has the prevalence of overweight, obesity and central obesity levelled off in the United States? Trends, patterns, disparities, and future projections for the obesity epidemic. Int J Epidemiol. 2020 Jun 1;49(3):810-823. doi: 10.1093/ije/dyz273. PMID 32016289
- [Background] Ogden CL, Fryar CD, Martin CB, Freedman DS, Carroll MD, Gu Q, Hales CM. Trends in Obesity Prevalence by Race and Hispanic Origin-1999-2000 to 2017-2018. JAMA. 2020 Sep 22;324(12):1208-1210. doi: 10.1001/jama.2020.14590. PMID 32857101
- [Background] McDow KB, Nguyen DT, Herrick KA, Akinbami LJ. Attempts to Lose Weight Among Adolescents Aged 16-19 in the United States, 2013-2016. NCHS Data Brief. 2019 Jul;(340):1-8. PMID 31442192
- [Background] Kakinami L, Houle-Johnson SA, Demissie Z, Santosa S, Fulton JE. Meeting fruit and vegetable consumption and physical activity recommendations among adolescents intending to lose weight. Prev Med Rep. 2018 Oct 28;13:11-15. doi: 10.1016/j.pmedr.2018.10.021. eCollection 2019 Mar. PMID 30456053
- [Background] Lucchini M, O'Brien LM, Kahn LG, Brennan PA, Glazer Baron K, Knapp EA, Lugo-Candelas C, Shuffrey L, Dunietz GL, Zhu Y, Wright RJ, Wright RO, Duarte C, Karagas MR, Ngai P, O'Connor TG, Herbstman JB, Dioni S, Singh AM, Alcantara C, Fifer WP, Elliott AJ; Environmental influences on Child Health Outcomes. Racial/ethnic disparities in subjective sleep duration, sleep quality, and sleep disturbances during pregnancy: an ECHO study. Sleep. 2022 Sep 8;45(9):zsac075. doi: 10.1093/sleep/zsac075. PMID 35724979
- [Background] Alves JM, Chow T, Nguyen-Rodriguez S, Angelo B, Defendis A, Luo S, Smith A, Yunker AG, Xiang AH, Page KA. Associations Between Sleep and Metabolic Outcomes in Preadolescent Children. J Endocr Soc. 2022 Sep 19;6(11):bvac137. doi: 10.1210/jendso/bvac137. eCollection 2022 Oct 11. PMID 36249413
- [Background] Okoli A, Hanlon EC, Brady MJ. The Relationship between Sleep, Obesity, and Metabolic Health in Adolescents - a Review. Curr Opin Endocr Metab Res. 2021 Apr;17:15-19. doi: 10.1016/j.coemr.2020.10.007. Epub 2020 Nov 4. PMID 33283071
- [Background] Weiss A, Xu F, Storfer-Isser A, Thomas A, Ievers-Landis CE, Redline S. The association of sleep duration with adolescents' fat and carbohydrate consumption. Sleep. 2010 Sep;33(9):1201-9. doi: 10.1093/sleep/33.9.1201. PMID 20857867
- [Background] Wilfley DE, Kass AE, Kolko RP. Counseling and behavior change in pediatric obesity. Pediatr Clin North Am. 2011 Dec;58(6):1403-24, x. doi: 10.1016/j.pcl.2011.09.014. PMID 22093859
- [Background] Dicker D, Alfadda AA, Coutinho W, Cuevas A, Halford JCG, Hughes CA, Iwabu M, Kang JH, Nawar R, Reynoso R, Rhee N, Rigas G, Salvador J, Sbraccia P, Vazquez-Velazquez V, Caterson ID. Patient motivation to lose weight: Importance of healthcare professional support, goals and self-efficacy. Eur J Intern Med. 2021 Sep;91:10-16. doi: 10.1016/j.ejim.2021.01.019. Epub 2021 Feb 6. PMID 33558163
- [Background] Coppell KJ, Abel SL, Freer T, Gray A, Sharp K, Norton JK, Spedding T, Ward L, Whitehead LC. The effectiveness of a primary care nursing-led dietary intervention for prediabetes: a mixed methods pilot study. BMC Fam Pract. 2017 Dec 21;18(1):106. doi: 10.1186/s12875-017-0671-8. PMID 29268719
- [Background] Mitchell TB, Amaro CM, Steele RG. Pediatric weight management interventions in primary care settings: A meta-analysis. Health Psychol. 2016 Jul;35(7):704-713. doi: 10.1037/hea0000381. Epub 2016 Apr 18. PMID 27089458
- [Background] Channon SJ, Huws-Thomas MV, Rollnick S, Hood K, Cannings-John RL, Rogers C, Gregory JW. A multicenter randomized controlled trial of motivational interviewing in teenagers with diabetes. Diabetes Care. 2007 Jun;30(6):1390-5. doi: 10.2337/dc06-2260. Epub 2007 Mar 10. PMID 17351283
- [Background] Beals E, Deierlein A, Katzow M. Clinical interventions to increase vegetable intake in children. Curr Opin Pediatr. 2023 Feb 1;35(1):138-146. doi: 10.1097/MOP.0000000000001203. Epub 2022 Nov 17. PMID 36385196
- [Background] DeBar LL, Stevens VJ, Perrin N, Wu P, Pearson J, Yarborough BJ, Dickerson J, Lynch F. A primary care-based, multicomponent lifestyle intervention for overweight adolescent females. Pediatrics. 2012 Mar;129(3):e611-20. doi: 10.1542/peds.2011-0863. Epub 2012 Feb 13. PMID 22331335
- [Background] Tucker SJ, Ytterberg KL, Lenoch LM, Schmit TL, Mucha DI, Wooten JA, Lohse CM, Austin CM, Mongeon Wahlen KJ. Reducing pediatric overweight: nurse-delivered motivational interviewing in primary care. J Pediatr Nurs. 2013 Nov-Dec;28(6):536-47. doi: 10.1016/j.pedn.2013.02.031. Epub 2013 Mar 24. PMID 23531463